CLINICAL TRIAL: NCT02561858
Title: Toxicity of Perirenal Fat in Overweight or Obese Subjects: A Pathophysiological Link Between Uric Acid Stones and Renal Ammonium Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-AOI-07
Record Dates: First submitted 2015-09-22; First posted 2015-09-28 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Uric Acid Stones
Keywords: Renal Ammonium ;uric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acid load test (Experimental)
  Interventions: Other: acid load test

INTERVENTIONS:
Other: acid load test

SUMMARY:
Patients who are overweight or obese, diabetic or not, share with those who are suffering from uric stones the same way to remove abnormal acidity of the body in urine, ie a kidney ammoniogenesis default. This results in an overly acidic urine pH which is directly pathogenic in people predisposed to develop uric stones because the precipitation of urate soluble uric acid is accelerated in acid medium.

Excess visceral fat, particularly perirenal, this defect may promote formation of renal ammonium. Indeed, the perirenal fat is adjacent to the renal cortex and shares with it a common arterial supply via the plexus Turner. Adipokines and fatty acids of the perirenal fat are predisposed to gain the renal cortex, seat of the ammoniogenesis. In humans the pathogenic role of the perirenal fat is demonstrated in chronic kidney disease and essential hypertension. However, the amount of fat and perirenal that of intra-abdominal fat are positively correlated.

Investigators hypothesis is that the perirenal fat also exert a pathogenic role in uric because of anatomical links between kidney stones and greasy environment and because excess fatty acids reaching the renal cortex decreases ammoniogenesis in an animal model metabolic syndrome.

For the test, the investigators will compare the amount of fat and perirenal renal ability to form ammonium in patients with uric or calcium lithiasis taking into account the amount of intra-abdominal fat.

ELIGIBILITY:
Inclusion Criteria:

* Urolithiasis Uric defined by more than 90% of uric acid anhydrous and / or dihydrate or calcium lithiasis defined by more than 90% mono calcium oxalate and / or dihydrate, and / or carbapatite and / or brushite;
* Overweight and obesity defined by 25 <BMI <35 kg / m2

Exclusion Criteria:

* staghorn lithiasis, stones struvite or cystine;
* Primary hyperparathyroidism;
* Hyperthyroidism;
* Any form of calcium or uric lithiasis secondary;
* Abnormal kidney structure (cysts, cortical thinning, kidney tumor);

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
the perirenal fat thickness (left) | baseline
  This is the perirenal fat thickness measured between the left posterior wall of the kidney and the posterior wall of the abdominal cavity on a TDM section in the plane of the left renal vein.

SECONDARY OUTCOMES:
the perirenal fat thickness (right) | baseline
  the average thickness of perirenal fat measured to the right
NH4 + / NAE | at day 7 of a standard diet
  It is the ratio NH4 + / NAE measured over 24 hours of urine collected at day 7 of a standard diet; it determines from acid removed as ammonium whose production is regulated physiologically by the kidneys
net acid urinary flow | at day 7 of a standard diet and when urine pH became <5.5
  This is the net acid urinary flow and report NH4 + / creat obtained when the urine pH became <5.5, in an acidic filler.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France